CLINICAL TRIAL: NCT03329495
Title: A Randomized Controlled Clinical Trial to Investigate the Effect of SMA- or SMV- Orientated Laparoscopic Right Hemicoloectomy for Right Colon Cancer With a Medial-to-lateral Approach
Brief Title: Laparoscopic Right Hemicoloectomy for Right Colon Cancer With a Medial-to-lateral Approach Orientated by SMA or SMV
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRSYM201710
Record Dates: First submitted 2017-10-30; First posted 2017-11-06 (Actual); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Right Colic Lymphadenopathy
Keywords: right colon cancer; superior mesenteric artery; superior mesenteric vein

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SMA-orientated right hemicoloectomy (Active Comparator): SMA-orientated right hemicoloectomy
  Interventions: Procedure: SMA-orientated right hemicoloectomy
- SMV-orientated right hemicoloectomy (Experimental): SMV-orientated right hemicoloectomy
  Interventions: Procedure: SMV-orientated right hemicoloectomy

INTERVENTIONS:
Procedure: SMA-orientated right hemicoloectomy — Laparoscopic right hemicoloectomy for right colon cancer with a medial-to-lateral approach orientated by SMA. The left boundary of resection is the left side of SMA, and artery sheath is not necessarily being opened.
  Arms: SMA-orientated right hemicoloectomy
Procedure: SMV-orientated right hemicoloectomy — Laparoscopic right hemicoloectomy for right colon cancer with a medial-to-lateral approach orientated by SMV. The left boundary of resection is the left side of SMV, and SMA is not exposed.
  Arms: SMV-orientated right hemicoloectomy

SUMMARY:
A randomized controlled clinical trial to compare the outcomes of SMA- and SMV- orientated laparoscopic right hemicoloectomy for right colon cancer with a medial-to-lateral approach

DETAILED DESCRIPTION:
In 2008, Germany scholar W. Hohenberger proposed the idea of complete mesocolic excision (CME) and central vascular ligation (CVL) for the standardization of colonic cancer surgery. This concept has been widely recognized and accepted. This radical operation attempts to remove the mesocolon intactly by careful dissection along the embryologic tissue planes and transection of the supplying vessels at their origin. For right-sided colon cancer, this approach involves division of the vessels at their origin from the superior mesenteric artery (SMA) and superior mesenteric vein (SMV). In our opinion, full exposure of the SMA and SMV is necessary to make sure that the origin of the colonic arteries being truly exposed and tied centrally at their origin and a maximal harvest of the regional lymphnodes. For locally advanced colon cancer, SMA- orientated surgery may be more meaningful to recerve a radical lymphadenectomy and bring benefit for their survival. However, in the traditional practise, the lymph node dissection is orientated by SMV and SMA is not exposed, tissue around SMA is left behind.

In this study, eligible patients with right colon cancer will be randomly allocated to receive either SMA- or SMV- orientated laparoscopic right hemicoloectomy. 100 patients will be enrolled in each group. In SMV- orientated surgery group, SMA is not exposed and the left boundary of resection is the left side of SMV. In SMA- orientated surgery group, the left boundary of resection is the left side of SMA and SMA is exposed.Artery sheath is not necessarily to be opened. Postoperative pathology will be analyzed with the number of lymph nodes retrieved. Postoperative recovery process and long term survival will be followed.

ELIGIBILITY:
Inclusion Criteria:

* Patients suitable for curative surgery between 18 - 85 years old;
* American Society of Anesthesiologists(ASA) grade I-III;
* Preoperative pathological diagnosis of adenocarcinoma;
* Tumor located at the right colon;
* Informed consent;
* No history of familial adenomatous polyposis, ulcerative colitis or Crohn's disease.

Exclusion Criteria:

* Pregnant patient;
* History of psychiatric disease;
* Use of systemic steroids;
* Simultaneous multiple primary colorectal cancer;
* Preoperative enhanced CT scan of chest, abdominal and pelvic cavity shows:

  1. Tumor involves the surrounding organs and combined organ resection needed to be done;
  2. distant metastasis;
  3. unable to perform R0 resection;
* History of any other malignant tumor in recent 5 years;
* Patients need emergency operation: mechanic ileus, perforation.
* Not suitable for laparoscopic surgery (i.e., extensive adhesion caused by abdominal surgery, not suitable for artificial pneumoperitoneum, etc).
* Conversion from laparoscopic surgery to laparotomy;

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2018-01 (Estimated); Primary Completion 2018-01 (Estimated); Study Completion 2023-01 (Estimated)

PRIMARY OUTCOMES:
number of lymph nodes retrieved | 1 day

SECONDARY OUTCOMES:
disease-free survival | 3 years
overall survival | 3 years
recurrence-free survival | 3 years
early complication rate | 30 days
  Early complication is defined as a complication that occurred between the finish of the surgery and postoperative day. Complications includes anastomotic leakage, anastomotic bleeding, chyle leakage, wound infection, pulmonary embolism, myocardial infarction et al.The Clavien-Dindo Classification of Surgical Complications will be applied to access the degree of severity of postoperative complications.
operative time | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Fumin Zhang, Professor, Principal Investigator — Ethics Committee of the First Affiliated Hospital, Nanjing Medical University, Jiangsu Province Hospital
Locations (1):
- Jiangsu province hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided